CLINICAL TRIAL: NCT00003392
Title: Multiple Cycles of High Dose Chemotherapy Supported With Filgrastim and Peripheral Blood Progenitor Cells in Patients With Metastatic Breast Cancer
Brief Title: High-Dose Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Recurrent or Refractory Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 9727; UNC-LCCC-970135 (Other: UNC IRB); NCI-G98-1446 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Melphalan; Paclitaxel; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim — 10 mcg/kg/d, day 2 through last day of leukapheresis
Drug: carboplatin — 18 AUC IV, approximately days 21, 42
Drug: cyclophosphamide — 4 gm/m2 IV, day 1
Drug: melphalan — 140 mg/m2 IV , approximately day 63
Drug: paclitaxel — 170 mg/m2 IV day 1
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of high-dose chemotherapy and peripheral stem cell transplantation in treating patients with recurrent or refractory metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effects on 2 year progression-free survival of a regimen consisting of cyclophosphamide, paclitaxel, and filgrastim (G-CSF) to mobilize peripheral blood progenitor cells (PBPCs), followed by 2 courses of carboplatin and paclitaxel followed by 1 course of melphalan, each supported with PBPCs and G-CSF, in patients with recurrent or refractory, advanced breast cancer. II. Evaluate the feasibility of administering multiple courses of high dose chemotherapy in an outpatient setting for these patients. III. Evaluate the rate of complete response to the high dose therapy in these patients.

OUTLINE: This is a multicenter study. Patients receive mobilization therapy consisting of cyclophosphamide IV over 1 hour followed by paclitaxel IV over 3 hours, then filgrastim (G-CSF) beginning 24 hours following completion of paclitaxel and continuing through the last day of leukapheresis. Leukapheresis continues until an adequate number of CD34+ cells is collected. Following cell count recovery, patients receive 3 courses of high-dose chemotherapy: 2 courses of paclitaxel IV over 3 hours followed by carboplatin IV over 1 hour, with the first course generally within 21 days after completion of leukapheresis and the second course 21-35 days after the first; then 1 course of melphalan IV infused over 30 minutes 21-35 days after the previous carboplatin dose. Each course of chemotherapy is followed 24-48 hours later by the infusion of G-CSF-mobilized peripheral blood progenitor cells and G-CSF. Patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 96 evaluable patients will be accrued for this study over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or refractory, metastatic breast cancer Patients previously treated for metastatic disease must show response to last standard dose chemotherapy regimen within 60 days of study entry OR Patients with no evidence of disease (e.g., resected skin lesions) must show no evidence of progression or bone disease No CNS metastases No disease progression following prior platinum or paclitaxel based regimens Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 to 65 Sex: Not specified Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 90,000/mm3 No prior inability to mobilize adequate peripheral blood progenitor cells for high dose therapy Hepatic: Bilirubin no greater than 1.8 mg/dL Transaminases stable and no greater than 3 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: LVEF within normal limits No significant cardiovascular disease No coronary artery disease No arrhythmias No congestive heart failure Other: Not pregnant or nursing Negative pregnancy test required of fertile women Effective contraception required of fertile patients Not HIV positive No nonmalignant disease precluding protocol treatment No sensitivity to E. coli-derived drug preparations No prior participation in this study No greater than grade I neurotoxicity

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior cellular support for high dose chemotherapy Chemotherapy: See Disease Characteristics No more than 6 prior courses of chemotherapy for metastatic disease At least 3 weeks since prior chemotherapy and recovered No prior high dose chemotherapy with cellular support Endocrine therapy: No concurrent steroid therapy Concurrent hormonal therapy allowed Radiotherapy: At least 3 weeks since prior radiotherapy and recovered No prior extensive pelvic radiation Surgery: Not specified Other: Recovered from acute toxic effects of any prior therapy No concurrent anticoagulation therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 1997-09; Primary Completion 2002-08 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Shea, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (14):
- United States (14):
  - Scripps Clinic, La Jolla, California
  - University of California San Diego, La Jolla, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Bone Marrow Stem Cell Transplant Institute of Florida, Fort Lauderdale, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Stem Cell Sciences, New York, New York
  - University of Rochester School of Medicine, Rochester, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Temple University Cancer Center, Philadelphia, Pennsylvania
  - Methodist Hospital-Central Unit, Memphis, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin